CLINICAL TRIAL: NCT04045665
Title: Anticoagulation for New-Onset Post-Operative Atrial Fibrillation After CABG
Acronym: PACES
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Annetine Gelijns, Chair, Department of Population Health Science & Policy Edmond A. Guggenheim Professor of Health Policy Co-Director, InCHOIR, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 08-1078; 2U01HL088942-12 (NIH)
Record Dates: First submitted 2019-08-02; First posted 2019-08-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Stroke; Bleeding
Keywords: Anticoagulation; Antiplatelet Therapy; Post Operative Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage | interventions — Anticoagulants

STUDY DESIGN:
Intervention Model Description: This is a multicenter randomized clinical trial comparing OAC to no-OAC in addition to concomitant antiplatelet therapy in 3,200 eligible patients who develop POAF after isolated CABG. The trial will be conducted by the Cardiothoracic Surgical Trials Network (CTSN), the German Society for Thoracic and Cardiovascular Surgery (DGTHG) and other European sites, the United Kingdom and Brazil..
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Antiplatelet Therapy (Active Comparator): Antiplatelet-only strategy
  Interventions: Drug: Antiplatelet-only strategy
- Oral Anticoagulant (Active Comparator): OAC-based strategy
  Interventions: Drug: Oral Anticoagulant plus background antiplatelet therapy

INTERVENTIONS:
Drug: Antiplatelet-only strategy — Aspirin 75-325 mg once-daily or a P2Y12-inhibitor (clopidogrel or ticagrelor)
  Arms: Antiplatelet Therapy
Drug: Oral Anticoagulant plus background antiplatelet therapy — OAC with vitamin K antagonist (VKA) with international normalized ratio (INR) target 2-3 or any approved direct oral anticoagulant OR apixaban, rivaroxaban, edoxaban or dabigatran) in addition to background antiplatelet therapy with aspirin 75-325mg once-daily or a P2Y12-inhibitor (clopidogrel or ticagrelor)
  Arms: Oral Anticoagulant

SUMMARY:
The primary objective of this study is to evaluate the effectiveness (prevention of thromboembolic events) and safety (major bleeding) of adding oral anticoagulation (OAC) to background antiplatelet therapy in patients who develop new-onset post-operative atrial fibrillation (POAF) after isolated coronary artery bypass graft (CABG) surgery.

All patients with a qualifying POAF event, who decline randomization, will be offered the option of enrollment in a parallel registry that captures their baseline risk profile and their treatment strategy in terms of anticoagulants or antiplatelets received. These patients will also be asked to fill out a brief decliner survey.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, randomized trial comparing OAC with no OAC (1:1 ratio) in patients who develop new-onset POAF after CABG. The primary effectiveness endpoint is the composite of death, ischemic stroke, transient ischemic attack (TIA), myocardial infarction (MI), systemic arterial thromboembolism or venous thromboembolism (VTE) at 90 days after randomization. The primary safety endpoint is BARC (Bleeding Academic Research Consortium) grade 3 or 5 bleeding at 90 days after randomization. The overall intent is to evaluate the trade-off in prevention of thromboembolic events versus an increase in bleeding.

Patients will be randomly assigned to the following treatment strategies:

* OAC-based strategy (experimental arm): OAC with vitamin K antagonist (VKA) with international normalized ratio (INR) target 2-3 or any approved direct oral anticoagulant (apixaban, rivaroxaban, edoxaban or dabigatran) in addition to background antiplatelet therapy with aspirin 75-325mg once-daily or a P2Y12-inhibitor (clopidogrel or ticagrelor)
* Antiplatelet-only strategy (control arm): single antiplatelet therapy with aspirin 75-325mg once-daily or a P2Y12-inhibitor (clopidogrel or ticagrelor)

The protocol-specified duration of anticoagulation is 90 days. Patients, who are randomized to the control arm and develop recurrent AF after 30 days, may be crossed-over to an OAC. Accrual is expected to take 60 months. Study follow-up visits will be performed at 90 days and phone follow-up at days 30, 60, and 180 days.

Data for patients enrolled in the registry will be ascertained from the local clinical site via a review of medical records. The baseline risk profile of registry patients (i.e., patients eligible but unwilling to be randomized) will be analyzed and compared to that of patients randomized in the trial. The usage of anticoagulant and antiplatelet therapies in the registry population overall and baseline CHA2DS2-VASC ischemic stroke risk score will also be determined.

Up to 500 patients will also be offered the option to participate in a digital health substudy which includes a wearable heart rhythm monitor device for 30 days post discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age ≥18 years who undergo isolated CABG for coronary artery disease
* POAF that persists for >60 minutes or is recurrent (more than one episode) within 7 days after the index CABG surgery

Exclusion Criteria:

* Clinical history of either permanent, persistent or paroxysmal atrial fibrillation
* Any pre-existing clinical indication for long-term OAC
* Any absolute contraindication to OAC
* Planned use of post-operative dual antiplatelet therapy (DAPT)

  a. This includes, but is not limited to, patients with recent PCI with drug-eluting or bare-metal stent.
* Cardiogenic shock
* Major perioperative complication* occurring between CABG and randomization

  a. including, but not limited to, stroke, TIA, MI, major bleeding (BARC type 4 bleeding), severe sepsis, renal failure requiring dialysis, or need for reoperation due to bleeding (e.g. pericardial tamponade).
* Concomitant left atrial appendage closure during CABG
* Concomitant valve surgery during CABG or prior valve surgery (including aortic, mitral, tricuspid or pulmonary)
* Concomitant mitral valve annuloplasty during CABG
* Concomitant carotid artery endarterectomy during CABG
* Concomitant aortic root replacement during CABG
* Concomitant surgery for AF during CABG
* Liver cirrhosis or Child-Pugh Class C chronic liver disease
* Pharmacologic therapy with an investigational drug or device within 30-days prior to randomization or plan to enroll patient in an investigational drug or device trial during participation in this trial
* Pregnancy at the time of randomization
* Unable or unwilling to provide inform consent
* Unable or unwilling to comply with the study treatment and follow-up
* Existence of underlying disease that limits life expectancy to less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Composite of death, ischemic stroke, TIA, MI, systemic arterial thromboembolism or venous thromboembolism (DVT and/or PE) | up to 180 days after randomization
  Composite score of death, ischemic stroke, transient ischemic attack (TIA), myocardial infarction (MI), systemic arterial thromboembolism or venous thromboembolism (deep venous thrombosis and/or pulmonary embolism). Composite score calculated by number of events.
Any BARC type 3 or 5 | 90 days after randomization
  The Bleeding Academic Research Consortium (BARC) - any type 3 or 5 bleeding thrombosis and/or pulmonary.
  Type 3: a. Overt bleeding plus hemoglobin drop of 3 to < 5 g/dL (provided hemoglobin drop is related to bleed); transfusion with overt bleeding
  b. Overt bleeding plus hemoglobin drop < 5 g/dL (provided hemoglobin drop is related to bleed); cardiac tamponade; bleeding requiring surgical intervention for control; bleeding requiring IV vasoactive agents
  c. Intracranial hemorrhage confirmed by autopsy, imaging, or lumbar puncture; intraocular bleed compromising vision.
  type 5: a. Probable fatal bleeding
  b. Definite fatal bleeding (overt or autopsy or imaging confirmation)

SECONDARY OUTCOMES:
Net clinical benefit (NCB) | 90 days after randomization
  Defined as the integration of the trial's primary effectiveness and safety endpoint to capture overall risk and benefit of anticoagulation. NCB will be assessed as a two-dimensional outcome with the observed NCB plotted versus effectiveness and safety, and a curve drawn. the confidence intervals will be compared to this curve.
Number of participants with Ischemic Stroke event | 180 days after randomization
Number of participants with TIA event | 180 days after randomization
Number of participants with MI event | 180 days after randomization
Number of participants with systematic arterial thromboembolism event | 180 days after randomization
Number of participants with venous thromboembolism event | 180 days after randomization
Number of cardiovascular mortalities | up to 180 days after randomization
Number of non-cardiovascular mortalities | up to 180 days after randomization
The incidence of BARC 2 bleeding at 90 after randomization | 90 days after randomization
  BARC Type 2: Any clinically overt sign of hemorrhage that "is actionable" and requires diagnostic studies, hospitalization, or treatment by a health care professional
The incidence of BARC 2 bleeding at 180 days after randomization | 180 days after randomization
  BARC Type 2: Any clinically overt sign of hemorrhage that "is actionable" and requires diagnostic studies, hospitalization, or treatment by a health care professional
Number of cardiac arrhythmias | 180 days after randomization
  Number of cardiac arrhythmias including recurrent symptomatic or asymptomatic AF requiring medical attention

CONTACTS AND LOCATIONS:
Overall Officials: Annetine C Gelijns, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Marc Gillinov, MD, Study Director — The Cleveland Clinic; John Alexander, MD, Study Director — Duke University
Locations (101):
- United States (51):
  - CHI St. Vincent, Arkansas, Little Rock, Arkansas
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - Medical Center of Aurora, Aurora, Colorado
  - Western Connecticut Hospital Systems, Danbury, Connecticut
  - Yale Medicine, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Piedmont Healthcare Inc., Atlanta, Georgia
  - Lutheran Medical Center, Fort Wayne, Indiana
  - Indiana University, Indianapolis, Indiana
  - Ascension St. Vincent, Indianapolis, Indiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Baystate Health, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Mid America Health Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Northwell Health System, Great Neck, New York
  - The Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - WakeMed, Raleigh, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Ascension St. John, Tulsa, Oklahoma
  - University of Pittsburgh Medical Center, Hermitage, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - Baylor Research Institute, Plano, Texas
  - Intermountain CV Research, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Health, Falls Church, Virginia
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
- Canada (9):
  - University of Alberta Hospital, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - University of Ottawa Heart Institute, Ottawa
  - Hôpital Laval, Québec
  - Toronto General Hospital, Toronto
- Germany (25):
  - University Heart Center Hamburg, Berlin, Brandenburg
  - Heart Center Leipzig, Berlin, Brandenburg
  - University Medical Center Göttingen, Göttingen, Lower Saxony
  - University Medical Center Jena, Jena, Thuringia
  - Kerckhoff Klinik, Bad Nauheim, Bad Nauheim
  - Clinic Bad Neustadt - Medical Center for Heart and Vascular Diseases, Bad Neustadt an der Saale
  - HDZ-NRW Bad Oeynhausen, Bad Oeynhausen
  - Charité Berlin - Benjamin Franklin Campus, Berlin
  - Charité Berlin - Rudolf Virchow Campus, Berlin
  - German Heart Center Berlin, Berlin
  - University Hospital Bonn, Bonn
  - Medical Center Braunschweig, Braunschweig
  - Heinrich Heine University Düsseldorf, Düsseldorf
  - Frankfurt University Hospital, Frankfurt
  - University Medical Center Frankfurt, Frankfurt
  - Heart Center, University of Freiburg, Freiburg im Breisgau
  - University Medical Center Halle, Halle
  - University Medical Center Heidelberg, Heidelberg
  - University Medical Center Schleswig-Holstein Kiel, Kiel
  - University Medical Center Schleswig-Holstein Lübeck, Lübeck
  - University Hospital Magdeburg, Magdeburg
  - German Heart Center Munich, Munich
  - Medical Center of the Ludwig-Maximilians-University Munich, Munich
  - University of Oldenburg, Oldenburg
  - Hospital of the Brothers of Mercy Trier, Trier
- United Kingdom (16):
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool, England
  - Barts Health NHS Trust, London, England
  - Imperial College Healthcare NHS Trust, London, England
  - Royal Wolverhampton NHS Trust, Wolverhampton, England
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Hull University Teaching Hospitals NHS Trust, Cottingham
  - University Hospitals of Leicester NHS Trust, Leicester
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - University Hospitals Sussex NHS Foundation Trust, Worthing

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: OtherDe-identified study data sets must be submitted to the designated NHLBI Program Official no later than 3 years after the end of the clinical activity (final patient follow-up, etc.) or 2 years after the main paper of the trial has been published, whichever comes first. Data are prepared by the study coordinating center and sent to the designated PO for review prior to release.
Access Criteria: Anyone who wishes to access the data.Any purpose.Data are available indefinitely at (Link to be included).
URL: https://biolincc.nhlbi.nih.gov/studies/

REFERENCES:
- [Derived] Budd AN, Kertai MD, Wyler von Ballmoos MC, Raphael J, Ghadimi K, Levy JH, Shore-Lesserson LJ, Mazzeffi MA, Sniecinski RM, Tanaka KA, Bolliger D, Abdalla M, Ural KG, Upchurch PA, Rozental O, Hunter CB, Seibert AR, Klick JC, Carroll D, Lobner K, Hensley NB. Management of Direct Oral Anticoagulants in Adult Patients Undergoing Cardiac Surgery: A Joint Consensus Statement by the Society of Cardiovascular Anesthesiologists and the Society of Thoracic Surgeons. Anesth Analg. 2026 Jan 29. doi: 10.1213/ANE.0000000000007868. Online ahead of print. PMID 41609362
- [Derived] Taha A, Nielsen SJ, Bergfeldt L, Ahlsson A, Friberg L, Bjorck S, Franzen S, Jeppsson A. New-Onset Atrial Fibrillation After Coronary Artery Bypass Grafting and Long-Term Outcome: A Population-Based Nationwide Study From the SWEDEHEART Registry. J Am Heart Assoc. 2021 Jan 5;10(1):e017966. doi: 10.1161/JAHA.120.017966. Epub 2020 Nov 30. PMID 33251914
- See also: The Cardiothoracic Surgical Trials Network — http://www.ctsurgerynet.org/index.html